CLINICAL TRIAL: NCT02174445
Title: Imatinib Continuation Versus Nilotinib 300 mg Twice Daily in Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase and Major Molecular Re-sponse (MMR) Without Molecular Response ≥ 4.5 Log (MR4.5) Receiving Imatinib at a Dose of 400 to 800 mg Daily. An Open-label, Randomised Multicenter Phase 3b Study to Determine the Confirmed Rate of Molecular Response ≥ 4 Log (MR4) at Two Years
Brief Title: An Open-label, Randomised Multicenter Phase 3b Study to Determine the Confirmed Rate of Molecular Response ≥ 4 Log (MR4) at Two Years
Acronym: DECLINE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: very slow recruitment rate and a lot of pat. didn't fulfil BCR-ABL requirements
Sponsor: Prof. Dr. Nikolas von Bubnoff (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Nikolas von Bubnoff, Mr., University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ADE18T; 2013-000077-68 (EudraCT Number); DRKS00006285 (Registry Identifier: DRKS)
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Patients with CML in chronic phase; Imatinib; Nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imatinib (Experimental): Imatinib 400-800mg, daily, maximum 6 years
  Interventions: Drug: Imatinib
- Nilotinib (Active Comparator): Nilotinib, 300mg, twice daily, maximum 6 years
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Imatinib — Imatinib, 400 to 800 mg p.o., daily
  Other Names: Glivec
  Arms: Imatinib
Drug: Nilotinib — 300mg p.o., twice-daily
  Other Names: Tasigna
  Arms: Nilotinib

SUMMARY:
This is an open-label, multicenter, randomised phase 3b clinical trial of Imatinib 400 to 800 mg daily versus Nilotinib 300 mg two times daily in chronic phase CML patients with confirmed MMR without MR4.5

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomised phase 3b clinical trial of Imatinib 400 to 800 mg daily versus Nilotinib 300 mg two times daily in chronic phase CML patients with confirmed MMR without MR4.5 (after having received Imatinib 400 to 800 mg daily for at least 18 months) to determine the proportion of patients with confirmed MR4 after two years. Patients in treatment arm A (Imatinib) who do not achieve confirmed MR4 2 years after randomisation will be offered cross-over from Imatinib 400 to 800 mg daily to Nilotinib 300 mg twice daily. One hundred thirty-two (132) patients will be included and randomised 1:1 to each treatment arm.

The study will be stratified by duration of Imatinib treatment before screen-ing (≤36 months / >36 months) as well as by the level of response at inclusion (MMR / MR4).

ELIGIBILITY:
Inclusion criteria:

1. Signed written informed consent
2. Male or female patients aged >=18 years (without upper limit of age)
3. ECOG performance status of 0 to 2
4. CML in chronic phase, with chronic phase defined as blasts < 15% in blood and/or bone marrow and peripheral blood basophils < 20% and platelets ≥ 100 G/L
5. Pretreatment with Imatinib with a treatment duration of at least 18 months at a dosage of 400 to 800 mg daily
6. Major molecular response (MMR) without molecular response ≥ 4.5 log (MR4.5), i.e. BCR-ABL>0.0032% and ≤0.1% IS confirmed by central la-boratory at screening will be required for randomisation
7. Patients must have a serum Creatinine of ≤ 1.5 x ULN, SGOT ≤ 1.5 x ULN, total bilirubin ≤ 1.5 x ULN (except known M. Gilbert), and Lipase ≤ 1.5 x ULN
8. Women of child-bearing potential defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months, must have a negative serum pregnancy test during screening period. Male and fe-male patients of reproductive potential must agree to employ highly ef-fective methods of birth control throughout the study and for up to 3 months following discontinuation of study drug. Appropriate methods are e.g. a highly effective method of first choice, i.e. a method with a low failure rate (less than 1% per year) like sexual abstinence, com-bined oral contraceptives, implants, injectable, some Intra Uterine Devices (IUDs), vasectomized partner, in combination with a method of second choice like condom, diaphragm, or cup pessary with spermicidal foam/gel/film/cream/suppository.

Exclusion Criteria:

1. Any previous treatment for CML other than Hydroxyurea, Imatinib or Interferon alpha
2. Evidence of features of accelerated or blast phase at any time
3. Previous loss of hematologic or cytogenetic response
4. Concomitant medications known to be strong inducers or inhibitors of P450 Isoenzyme CYP3A4
5. Finding of a secondary BCR-ABL resistance mutation at any time
6. History of intolerance to Imatinib that required treatment interruption longer than 4 weeks (cumulative) or dose reductions to less than 400 mg daily for longer than 4 weeks (cumulative) during the last 12 months before informed consent
7. Patients who had prior allogeneic, syngeneic, or autologous bone mar-row transplant or stem cell transplant
8. Patients unwilling to or unable to comply with the planned therapeutic intervention or to comply with the study treatment visits including blood sample collection within the protocol
9. History of pancreatitis, chronic inflammatory diseases or autoimmune diseases
10. Patients who underwent solid organ transplantation
11. Impaired cardiac function, including any of the following:

    * History of or presence of complete left bundle branch block, right bundle branch block plus left anterior hemi block, bifascicular block in screening ECG
    * Use of a cardiac pacemaker
    * ST depression of > 1mm in 2 or more leads and/or T wave inver-sions in 2 or more contiguous leads in screening ECG
    * Congenital Long QT Syndrome
    * QTc> 450 msec in the screening ECG
    * QT prolonging concomitant medication
    * History of or presence of significant ventricular or atrial tachy-arrhythmia in screening ECG
    * History of or presence of clinically significant resting bradycardia (< 50 beats per minute)
    * Myocardial infarction within 12 months prior to informed consent
    * Unstable angina diagnosed or treated during the past 12 months before informed consent
    * Other clinically significant heart disease (e.g., congestive heart fail-ure, uncontrolled hypertension, history of labile hypertension)
12. Known HIV and/or hepatitis B or C infection (testing is not mandatory)
13. Other malignancies within the past 3 years before informed consent except for adequately treated carcinoma of the cervix and basal or squamous cell carcinoma of the skin
14. Women who are pregnant or breast feeding
15. Male/female patients of reproductive potential unwilling to practice a highly effective method of birth control
16. History of noncompliance to medical regimens
17. Treatment with another investigational product during this study or during the last 30 days prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with confirmed MR4 after two years of study treatment | 2 years
  Proportion of patients with confirmed MR4 at two years of study treatment in both treatment arms. Confirmed MR4 at two years is defined as either BCR-ABL ≤ 0.01% IS at 21 and 24 months or BCR-ABL ≤ 0.01% IS at 24 months and confirmation within six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nikolas von Bubnoff, Professor, Principal Investigator — University Hospital Freiburg
Locations (18):
- Germany (18):
  - Universitätsklinikum Aachen, Aachen
  - Praxis Dr. Bruder / Dr. Heinrich / Prof. Bangerter, Augsburg
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinik Köln, Cologne
  - Gemeinschaftspraxis, Dresden
  - Praxis Dr. Hauch, Erfurt
  - Internistische Schwerpunktpraxis Erlangen oncosearch, Erlangen
  - Praxis für Hämatologie/Onkologie Dres. Rudolph, Sengpiel, von Verschuer, Essen
  - University Medical Center, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Gemeinschaftspraxis Hämatologie/Onkologie, Magdeburg
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Überörtliche Gemeinschaftspraxis Hämato-Onkologie Pasing/Fürstenfeldbruck, Munich
  - Klinikum rechts der Isar, Technische Universität München, München
  - Onkologische Praxis Oldenburg, Oldenburg
  - Medizinische Statistik Saarbrücken, GbR, Saarbrücken
  - Universitätsklinikum Ulm, Ulm